CLINICAL TRIAL: NCT00667446
Title: A 36 Month, Multi-Center, Open-Label Extension Study to Evaluate the Safety of Leuprolide Acetate 11.25 mg and 30 mg Formulations in Children With Central Precocious Puberty
Brief Title: Safety Extension Study Of Leuprolide Acetate (Lupron Depot) In The Treatment Of Central Precocious Puberty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-CP07-177
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Precocious; Leuprolide Acetate; Luteinizing Hormone (LH); Gonadotrophin-releasing Hormone Agonist (GnRHa); Tanner Staging; Depot Formulation; Suppression of LH; Central Precocious Puberty (CPP); Gonadotrophin-releasing Hormone (GnRH); Lupron; GnRH Analog; Pediatrics Central Precocious Puberty
Keywords: GnRH analog; Luteinizing hormone (LH); Gonadotrophin-releasing hormone agonist(GnRHa); Suppression of LH; Gonadotrophin-releasing hormone (GnRH); CPP; Leuprolide acetate; Central Precocious Puberty; Depot formulation; Lupron; Tanner staging; Pediatrics
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leuprolide Acetate 3M Depot 11.25 mg (Experimental): Twelve intramuscular injections of leuprolide acetate for depot suspension 11.25 mg administered 3 months (3M) apart.
  Interventions: Drug: Leuprolide Acetate 3 Month Depot
- Leuprolide Acetate 3M Depot 30 mg (Experimental): Twelve intramuscular injections of leuprolide acetate for depot suspension 30 mg administered 3 months apart.
  Interventions: Drug: Leuprolide Acetate 3 Month Depot

INTERVENTIONS:
Drug: Leuprolide Acetate 3 Month Depot
  Other Names: ABT-818; Lupron; Leuprorelin acetate

SUMMARY:
The purpose of this extension study is to determine if leuprolide acetate (11.25 mg and 30 mg) is safe in treating children with Central Precocious Puberty over a longer period of time (36 months).

DETAILED DESCRIPTION:
This study includes a 36-month Study Drug Treatment Period (3-month treatment cycles), and a Safety Follow-up Period (12 weeks following the Month 36 visit). Participants will receive a total of twelve injections of the same treatment they received in the lead-in study, L-CP07-167 (NCT00635817) either leuprolide acetate 11.25 mg or 30 mg depot formulation. Each injection will be administered 3 months apart for up to 36 months of treatment. Study visits will occur on Day 1, Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30 and 33 (1st through the 12th leuprolide acetate depot injections, respectively), Month 36, and 12 weeks later for the Safety Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the Treatment Period of the lead-in study, L-CP07-167 (NCT00635817), and has documented luteinizing hormone suppression as evidenced by peak-stimulated luteinizing hormone <4 mIU/mL at the Month 6 study visit of the lead-in study.
* Demonstrated suppression of the physical signs of puberty at Month 6 of the lead-in study.
* Subject is expected to receive at least 12 months of therapy to treat Central Precocious Puberty after study entry.
* In general good health with no uncontrolled, clinically significant disease which would interfere with bone maturation or mask the objectives of this protocol as assessed by the investigator.

Exclusion Criteria:

* Incomplete precocious puberty, peripheral precocious puberty or evidence of any abnormal pituitary, hypothalamic, adrenal, thyroid and gonadal function (other than premature secretion of gonadotropins) not adequately controlled, unstable intracranial tumors except hamartoma.
* Bone age ≥14 years for girls and ≥15 years for boys (based on the Month 6 lead in study, L-CP07-167, radiographic results).
* Has an abnormal laboratory value suggesting a clinically significant underlying disease or condition.
* Chronic illness requiring treatment that may interfere with growth, ie, chronic steroid use, renal failure, moderate to severe scoliosis.
* Current therapy with medroxyprogesterone acetate.
* Current therapy with growth hormone.
* Current therapy with insulin-like growth factor-1 (IGF-1).
* Current use of an estrogen preparation.
* Any concomitant medical condition that, in the opinion of the investigator, may expose a subject to an unacceptable level of safety risk or that affects subject compliance.
* Subject has a positive pregnancy test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-12; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bacher, MD, Study Director — AbbVie
Locations (20):
- United States (16):
  - Site Reference ID/Investigator# 13521, Birmingham, Alabama
  - Site Reference ID/Investigator# 14922, Long Beach, California
  - Site Reference ID/Investigator# 26043, Los Angeles, California
  - Site Reference ID/Investigator# 20802, San Diego, California
  - Site Reference ID/Investigator# 22425, Greenwood Village, Colorado
  - Site Reference ID/Investigator# 18181, Jacksonville, Florida
  - Site Reference ID/Investigator# 26364, Pensacola, Florida
  - Site Reference ID/Investigator# 26983, Indianapolis, Indiana
  - Site Reference ID/Investigator# 20821, Shreveport, Louisiana
  - Site Reference ID/Investigator# 23643, Minneapolis, Minnesota
  - Site Reference ID/Investigator# 23502, Saint Paul, Minnesota
  - Site Reference ID/Investigator# 14121, Kansas City, Missouri
  - Site Reference ID/Investigator# 23802, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 13324, Tulsa, Oklahoma
  - Site Reference ID/Investigator# 16506, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 14024, Seattle, Washington
- Puerto Rico (4):
  - Site Reference ID/Investigator# 23182, Bayamón
  - Site Reference ID/Investigator# 21721, Ponce
  - Site Reference ID/Investigator# 25908, Rio Piedras
  - Site Reference ID/Investigator# 23082, San Juan

REFERENCES:
- [Derived] Lee PA, Klein K, Mauras N, Lev-Vaisler T, Bacher P. 36-month treatment experience of two doses of leuprolide acetate 3-month depot for children with central precocious puberty. J Clin Endocrinol Metab. 2014 Sep;99(9):3153-9. doi: 10.1210/jc.2013-4471. Epub 2014 Jun 13. PMID 24926950
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who successfully completed and showed maintenance of luteinizing hormone suppression through the 6-month treatment period of the lead-in study L-CP07-167 (NCT00635817) received the same treatment in this study that they were previously assigned in the lead-in study.
Pre-assignment Details: At the end of the Treatment Period, participants who completed the study or prematurely discontinued from the study could enter the Safety Follow-Up Period.
Groups:
- Leuprolide Acetate 3M Depot 11.25 mg: Twelve intramuscular injections of leuprolide acetate for depot suspension 11.25 mg administered 3 months apart during the Treatment Period. During the Safety Follow-Up Period participants were offered standard of care treatment as deemed appropriate by the investigator.
- Leuprolide Acetate 3M Depot 30 mg: Twelve intramuscular injections of leuprolide acetate for depot suspension 30 mg administered 3 months apart during the Treatment Period. During the the Safety Follow-Up Period participants were offered standard of care treatment as deemed appropriate by the investigator.
Period: Treatment Period (36 Months)
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Started | 34 | 38
Completed | 11 | 13
Not Completed | 23 | 25
Not completed — Ready to enter puberty based on age | 13 | 15
Not completed — Other | 2 | 2
Not completed — Personal reasons | 2 | 2
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Not Adequately Suppressed on Therapy | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Therapeutic Failure | 1 | 1
Period: Safety Follow-up Period (12 Weeks)
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Started | 28 | 26
Completed | 28 | 25
Not Completed | 0 | 1
Not completed — No Longer Needed Treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug in this extension study.
Groups:
- Leuprolide Acetate 3M Depot 11.25 mg: Twelve intramuscular injections of leuprolide acetate for depot suspension 11.25 mg administered 3 months apart.
- Total: Total of all reporting groups
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.50 (1.71) | 8.45 (1.52) | 8.47 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Suppression of Peak-Stimulated Luteinizing Hormone
Description: Luteinizing Hormone (LH) suppression is defined as peak-stimulated LH < 4 mIU/mL. Peak-stimulated LH refers to the maximum LH concentration measured 30 and 60 minutes after a gonadotropin-releasing hormone agonist (GnRHa) stimulation test. Participants who failed suppression at previous visit and prematurely discontinued were counted as having failed future visits also. Final visit is the participant's last visit closest to Month 36.
Time Frame: Day 1, Months 6, 12, 24, and 36
Population: Intention-to-treat, defined as patients who received at least 1 dose of study drug with at least 1 post-baseline measurement of any maintenance of suppression variable, & did not prematurely discontinue in the 1st 30 days due to inadequate suppression at Month 6 of the lead-in study. N= the number of patients with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 33 | 38
percentage of participants
  Day 1 [N= 32, 37] | 96.9 [83.78 to 99.92] | 100.0 [90.51 to 100.00]
  Month 6 [N=32, 36] | 93.8 [79.19 to 99.23] | 100.0 [90.26 to 100.00]
  Month 12 [N=31, 32] | 90.3 [74.25 to 97.96] | 96.9 [83.78 to 99.92]
  Month 24 [N=16, 18] | 87.5 [64.65 to 98.45] | 100.0 [81.47 to 100.00]
  Month 36 [N=9, 11] | 77.8 [39.99 to 97.19] | 100.0 [71.51 to 100.00]
  Final Visit [N=33, 36] | 93.9 [79.77 to 99.26] | 100.0 [90.26 to 100.00]

2. Secondary Outcome: Percentage of Female Participants With Suppression of Basal Estradiol (Assay 1)
Description: The percentage of female participants with suppression of basal estradiol to prepubertal levels, defined as estradiol < 20 pg/mL.
  The estradiol assay was changed in June of 2010, and the lower limit of quantitation (LLOQ) was increased from 1 pg/mL to 10 pg/mL. This outcome measure reports data for assays performed before this change occurred, with an LLOQ of 1 pg/mL. Final visit is the participant's last visit closest to Month 36.
Time Frame: Day 1, Months 3, 6, 9, 12, and 24
Population: Intention-to-treat female population. N = the number of participants with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 31 | 33
percentage of participants
  Day 1 [N=28, 30] | 96.4 [81.65 to 99.91] | 100.0 [88.43 to 100.00]
  Month 3 [N=29, 33] | 100.0 [88.06 to 100.00] | 100.0 [89.42 to 100.00]
  Month 6 [N=26, 25] | 100.0 [86.77 to 100.00] | 100.0 [86.28 to 100.00]
  Month 9 [N=18, 18] | 100.0 [81.47 to 100.00] | 100.0 [81.47 to 100.00]
  Month 12 [N=10, 12] | 100.0 [69.15 to 100.00] | 100.0 [73.54 to 100.00]
  Month 24 [N=1, 0] | 100.0 [2.50 to 100.00] | NA [NA to NA] — No participants with available data at this time point
  Final Visit [N=31, 33] | 100.0 [88.78 to 100.00] | 100.0 [89.42 to 100.00]

3. Secondary Outcome: Percentage of Female Participants With Suppression of Basal Estradiol (Assay 2)
Description: The percentage of female participants with suppression of basal estradiol to prepubertal levels, defined as estradiol < 20 pg/mL.
  The estradiol assay was changed in June of 2010, and the lower limit of quantitation (LLOQ) was increased from 1 pg/mL to 10 pg/mL. This outcome measure reports data for assays performed after this change occurred, with an LLOQ of 10 pg/mL. Final visit is the participant's last visit closest to Month 36.
Time Frame: Months 6, 9, 12, 24, 30, and 36
Population: Intention-to-treat female population. N = the number of participants with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 31 | 33
percentage of participants
  Month 6 [N=4, 6] | 100.0 [39.76 to 100.00] | 83.3 [35.88 to 99.58]
  Month 9 [N=13, 10] | 61.5 [31.58 to 86.14] | 40.0 [12.16 to 73.76]
  Month 12 [N=20, 15] | 45.0 [23.06 to 68.47] | 60.0 [32.29 to 83.66]
  Month 24 [N=14, 15] | 50.0 [23.04 to 76.96] | 53.3 [26.59 to 78.73]
  Month 30 [N=9, 15] | 33.3 [7.49 to 70.07] | 26.7 [7.79 to 55.10]
  Month 36 [N=7, 11] | 28.6 [3.67 to 70.96] | 36.4 [10.93 to 69.21]
  Final Visit [N=24, 26] | 29.2 [12.62 to 51.09] | 30.8 [14.33 to 51.79]

4. Secondary Outcome: Percentage of Male Participants With Suppression of Basal Testosterone
Description: The percentage of male participants with suppression of basal testosterone to prepubertal levels, defined as testosterone < 30 ng/dL. Final visit is the participant's last visit closest to Month 36.
Time Frame: Day 1, Months 3, 6, 9, 12, 24, 30, and 36
Population: Intention-to-treat male population. N = the number of participants with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 2 | 5
percentage of participants
  Day 1 [N= 2, 5] | 100.0 [15.81 to 100.00] | 100.0 [47.82 to 100.00]
  Month 3 [N=2, 5] | 100.0 [15.81 to 100.00] | 100.0 [47.82 to 100.00]
  Month 6 [N=2, 5] | 100.0 [15.81 to 100.00] | 80.0 [28.36 to 99.49]
  Month 9 [N=2, 5] | 100.0 [15.81 to 100.00] | 80.0 [28.36 to 99.49]
  Month 12 [N=1, 5] | 100.0 [2.50 to 100.00] | 100.0 [47.82 to 100.00]
  Month 24 [N=1, 3] | 100.0 [2.50 to 100.00] | 66.7 [9.43 to 99.16]
  Month 30 [N=0, 1] | NA [NA to NA] — No participants with available data at this time point | 100.0 [2.50 to 100.00]
  Month 36 [N=0, 1] | NA [NA to NA] — No participants with available data at this time point | 100.0 [2.50 to 100.00]
  Final Visit [N=2, 5] | 100.0 [15.81 to 100.00] | 100.0 [47.82 to 100.00]

5. Secondary Outcome: Mean Peak-stimulated Luteinizing Hormone Concentration by Visit
Description: Peak-stimulated luteinizing hormone refers to the maximum luteinizing hormone concentration measured 30 and 60 minutes after a gonadotropin-releasing hormone agonist (GnRHa) stimulation test. Final visit is the participant's last visit closest to Month 36.
Time Frame: Baseline of the lead-in study L-CP07-167, Day 1, Months 6, 12, 24, and 36
Population: Intention-to-treat. N = the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 33 | 38
mIU/mL
  Baseline [N=33, 38] | 21.89 (38.46) | 10.16 (12.66)
  Day 1 [N=32, 37] | 2.00 (1.03) | 1.49 (0.86)
  Month 6 [N=32, 36] | 2.22 (1.16) | 1.62 (0.82)
  Month 12 [N=31, 32] | 2.24 (1.20) | 1.58 (1.02)
  Month 24 [N=14, 18] | 1.67 (0.97) | 0.88 (0.58)
  Month 36 [N=7, 11] | 1.51 (0.85) | 0.91 (0.49)
  Final Visit [N=33, 36] | 1.81 (1.13) | 1.15 (0.74)

6. Secondary Outcome: Percentage of Female Participants With Suppression of the Physical Signs of Puberty (Breast Development)
Description: The percentage of female participants with suppression of breast development. Breast development was rated from Stage 1 (early development) through Stage 5 (full development) according to a modified Tanner Staging pictogram. Suppression of breast development is defined as regression or no progression of breast development from Baseline (of the lead-in study L-CP07-167) according to pubertal staging. Girls entering the study with fully developed breasts (Stage 5) were excluded from this analysis. Final visit is the participant's last visit closest to Month 36.
Time Frame: Baseline (of the lead-in study L-CP07-167), Day 1, Months 3, 6, 9, 12, 18, 24, 30, and 36
Population: Intention-to-treat female population, excluding participants who entered the study at Stage 5. N = the number of participants with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 31 | 31
percentage of participants
  Day 1 [N= 31, 31] | 90.3 [74.2 to 98.0] | 83.9 [66.3 to 94.5]
  Month 3 [N=29, 31] | 86.2 [68.3 to 96.1] | 87.1 [70.2 to 96.4]
  Month 6 [N=31, 30] | 90.3 [74.2 to 98.0] | 80.0 [61.4 to 92.3]
  Month 9 [N=31, 28] | 87.1 [70.2 to 96.4] | 75.0 [55.1 to 89.3]
  Month 12 [N=28, 26] | 85.7 [67.3 to 96.0] | 80.8 [60.6 to 93.4]
  Month 18 [N=17, 20] | 82.4 [56.6 to 96.2] | 75.0 [50.9 to 91.3]
  Month 24 [N=14, 16] | 78.6 [49.2 to 95.3] | 75.0 [47.6 to 92.7]
  Month 30 [N=10, 16] | 90.0 [55.5 to 99.7] | 68.8 [41.3 to 89.0]
  Month 36 [N=8, 12] | 87.5 [47.3 to 99.7] | 66.7 [34.9 to 90.1]
  Final Visit [N=31, 31] | 83.9 [66.3 to 94.5] | 71.0 [52.0 to 85.8]

7. Secondary Outcome: Percentage of Male Participants With Suppression of the Physical Signs of Puberty (Testicular Volume and Genital Development)
Description: The percentage of male participants with suppression of testicular volume and genital staging. Testicular volume was calculated from the length, width and height of each testicle measured by ultrasound. External genital development (testes and penis) was rated from Stage 1 (early development) through Stage 5 (full development) according to a modified Tanner Staging pictogram. Suppression is defined as regression or no progression in both testicular volume and genital staging from Baseline (of the lead-in study L-CP07-167) according to pubertal staging. Boys entering the study with fully developed genitals (Stage 5) were excluded from this analysis. Final visit is the participant's last visit closest to Month 36.
Time Frame: Baseline (of the lead-in study L-CP07-167), Day 1, Months 3, 6, 9, 12, 18, 24, 30, and 36
Population: Intention-to-treat male population, excluding participants who entered the study at Stage 5. N = the number of participants with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 2 | 5
percentage of participants
  Day 1 [N= 2, 5] | 50.0 [1.3 to 98.7] | 40.0 [5.3 to 85.3]
  Month 3 [N=2, 5] | 50.0 [1.3 to 98.7] | 60.0 [14.7 to 94.7]
  Month 6 [N=2, 5] | 50.0 [1.3 to 98.7] | 60.0 [14.7 to 94.7]
  Month 9 [N=2, 5] | 50.0 [1.3 to 98.7] | 40.0 [5.3 to 85.3]
  Month 12 [N=1, 5] | 100.0 [2.5 to 100.0] | 60.0 [14.7 to 94.7]
  Month 18 [N=1, 3] | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0]
  Month 24 [N=1, 3] | 100.0 [2.5 to 100.0] | 33.3 [0.8 to 90.6]
  Month 30 [N=1, 1] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0]
  Month 36 [N=0, 1] | NA [NA to NA] — No participants with available data at this time point | 100.0 [2.5 to 100.0]
  Final Visit [N=2, 5] | 50.0 [1.3 to 98.7] | 20.0 [0.5 to 71.6]

8. Secondary Outcome: Change From Baseline in Growth Rate
Description: Baseline growth rate was the growth rate in the one year prior to Day 1 of the lead-in study L-CP07-167. Growth rates were calculated as the ratio of the change in height to the change in chronological age with an approximate 6-month interval for Day 1, Months 6, 12, 18, 24, 30, 36 and the Final Treatment Visit.
Time Frame: Baseline (the 1 year prior to the start of treatment in the lead-in study), and Day 1, Months 6, 12, 18, 24, 30, and 36
Population: Intention-to-treat with available growth rate data. N = participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 32 | 38
cm/year
  Baseline [N=32, 38] | 7.2 (3.96) | 7.53 (2.81)
  Change from Baseline at Day 1 [N=32, 38] | -1.67 (3.90) | -1.65 (3.43)
  Change from Baseline at Month 6 [N=32, 37] | -1.66 (3.78) | -2.04 (2.95)
  Change from Baseline at Month 12 [N=28, 32] | -1.99 (3.90) | -2.28 (2.88)
  Change from Baseline at Month 18 [N=18, 23] | -2.21 (4.29) | -2.06 (2.40)
  Change from Baseline at Month 24 [N=15, 19] | -2.36 (4.85) | -1.59 (2.20)
  Change from Baseline at Month 30 [N=11, 17] | -1.86 (5.45) | -2.13 (2.33)
  Change from Baseline at Month 36 [N=8, 13] | -2.64 (5.93) | -2.19 (2.41)
  Change from Baseline at Final Visit [N=32, 38] | -2.27 (3.78) | -2.64 (2.65)

9. Secondary Outcome: Ratio of Change From Baseline in Bone Age/Change From Baseline in Chronological Age
Description: Bone age was determined by left hand/wrist bone age radiographs that were evaluated using the Fels Method by a central reader. The ratio of change from Baseline in bone age (BA)/change from Baseline in chronological age (CA) was calculated using the following formula:
  (BA at Post-baseline Treatment Visit - BA at Baseline) / (CA at Post-baseline Treatment Visit - CA at Baseline).
Time Frame: Baseline (of the lead-in study L-CP07-167), and Day 1, Months 12, 24, and 36
Population: Intention-to-treat with available bone age data. N = participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Number analyzed (Participants) | 33 | 37
ratio
  Day 1 [N=32, 37] | 0.51 (0.56) | 1.02 (1.27)
  Month 12 [N=32, 32] | 0.52 (0.33) | 0.62 (0.37)
  Month 24 [N=14, 17] | 0.53 (0.30) | 0.72 (0.34)
  Month 36 [N=5, 11] | 0.43 (0.15) | 0.64 (0.30)
  Final Visit [N=33, 32] | 0.48 (0.28) | 0.56 (0.30)

ADVERSE EVENTS:
Time Frame: 37 months
Arm/Group | Leuprolide Acetate 3M Depot 11.25 mg | Leuprolide Acetate 3M Depot 30 mg
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/38
Other Adverse Events (participants affected / at risk) | 31/34 | 31/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate 3M Depot 11.25 mg (N=34) | Leuprolide Acetate 3M Depot 30 mg (N=38)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate 3M Depot 11.25 mg (N=34) | Leuprolide Acetate 3M Depot 30 mg (N=38)
EAR PAIN (Ear and labyrinth disorders) | 1 | 2
MYOPIA (Eye disorders) | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 3
CONSTIPATION (Gastrointestinal disorders) | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 3 | 2
NAUSEA (Gastrointestinal disorders) | 2 | 1
VOMITING (Gastrointestinal disorders) | 0 | 4
INJECTION SITE PAIN (General disorders) | 10 | 9
PYREXIA (General disorders) | 6 | 5
SEASONAL ALLERGY (Immune system disorders) | 2 | 1
BODY TINEA (Infections and infestations) | 3 | 0
BRONCHITIS (Infections and infestations) | 3 | 0
EAR INFECTION (Infections and infestations) | 3 | 1
GASTROENTERITIS (Infections and infestations) | 4 | 4
INFLUENZA (Infections and infestations) | 3 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 1
PHARYNGITIS (Infections and infestations) | 2 | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 5 | 4
SINUSITIS (Infections and infestations) | 2 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 | 5
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 2
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 2
WEIGHT INCREASED (Investigations) | 0 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 3
HEADACHE (Nervous system disorders) | 5 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 9
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 5
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
ACNE (Skin and subcutaneous tissue disorders) | 2 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 1
RASH (Skin and subcutaneous tissue disorders) | 3 | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.